CLINICAL TRIAL: NCT02765113
Title: Effect of Two Different Surgical Methods on the Prognosis of Patients With Blepharospasm
Brief Title: Two Different Surgical Methods of Blepharospasm
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-16-008
Record Dates: First submitted 2016-04-14; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-04

CONDITIONS: Blepharospasm
MeSH Terms: conditions — Blepharospasm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Facial nerve combing (Active Comparator): Facial nerve combing and Microvascular Decompression(MVD) was performed in all the patients in this group.
  Interventions: Procedure: Facial nerve combing
- Facial and Trigeminal nerve combing (Active Comparator): Facial nerve combing、trigeminal nerve combing and Microvascular Decompression(MVD) was performed in all the patients in this group.
  Interventions: Procedure: Facial and Trigeminal nerve combing

INTERVENTIONS:
Procedure: Facial nerve combing — Facial nerve combing:To sort out the facial nerve using the nerve combing knife.
  MVD: explore the facial nerve and trigeminal nerve and then perform microvascular decompression.
  Arms: Facial nerve combing
Procedure: Facial and Trigeminal nerve combing — Facial nerve combing:To sort out the facial nerve using the nerve combing knife.
  Trigeminal nerve combing:To sort out the trigeminal nerve using the nerve combing knife.
  MVD: explore the facial nerve and trigeminal nerve and then perform microvascular decompression.
  Arms: Facial and Trigeminal nerve combing

SUMMARY:
1. Background: Blepharospasm refers to orbital and periorbital orbicularis muscle spontaneous spasmodic contraction. Continuous spasm can be long or short, the performance of non spasm will strongly closed repeatedly. At present, the pathogenesis of blepharospasm is not clear, in addition, there is no particularly effective treatment.
2. Purpose：compare two different surgical methods, observe the improvement of symptoms and prognosis of patients with blepharospasm.
3. Scientific hypothesis: At present, the pathogenesis of blepharospasm is not clear, but clinical patients with blepharospasm showed bilateral eyelid twitching, eyes open difficulties and the symptoms are worse when tension, anxiety, insomnia, light stimulation and wind outside stimulation. At the same time, in the clinic，the investigators found that facial nerve and trigeminal nerve combing can improve the clinical symptoms of the patients. Therefore, the investigators speculated that over activity were related to clinical symptoms and corneal reflex pathway of blepharospasm patients.
4. Research content: the blepharospasm patients were randomly divided into two groups, prospective comparative analysis of two different surgical methods for the treatment of blepharospasm. One group of patients were performed facial nerve combing and microvascular decompression, the other group of patients were performed facial nerve, trigeminal nerve combing with microvascular decompression, to observation of postoperative clinical improvement of two groups of patients.
5. Expected results:To define a surgical method for the treatment of blepharospasm, and to promote the use of the academic and clinical practice.

DETAILED DESCRIPTION:
Background: Blepharospasm refers to orbital and periorbital orbicularis muscle spontaneous spasmodic contraction. Continuous spasm can be long or short, the performance of non spasm will strongly closed repeatedly. At present, the pathogenesis of blepharospasm is not clear, in addition, there is no particularly effective treatment.

Purpose：compare two different surgical methods, observe the improvement of symptoms and prognosis of patients with blepharospasm.

Scientific hypothesis: At present, the pathogenesis of blepharospasm is not clear, but clinical patients with blepharospasm showed bilateral eyelid twitching, eyes open difficulties and the symptoms are worse when tension, anxiety, insomnia, light stimulation and wind outside stimulation. At the same time, in the clinic，the investigators found that facial nerve and trigeminal nerve combing can improve the clinical symptoms of the patients. Therefore, the investigators speculated that over activity were related to clinical symptoms and corneal reflex pathway of blepharospasm patients.

Research content: the blepharospasm patients were randomly divided into two groups, prospective comparative analysis of two different surgical methods for the treatment of blepharospasm. One group of patients were performed facial nerve combing and microvascular decompression, the other group of patients were performed facial nerve, trigeminal nerve combing with microvascular decompression, to observation of postoperative clinical improvement of two groups of patients.

Expected results:To define a surgical method for the treatment of blepharospasm, and to promote the use of the academic and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bilateral blepharospasm
2. Clinical symptoms more than 1 years.
3. Patients who are willing to undergo surgery.
4. Preoperative patients who had not been treated with botulinum toxin.

Exclusion Criteria:

1. Patients with serious heart and lung dysfunction can not tolerate surgery.
2. The clinical symptoms of the patients less than 1 years.
3. Patients who received local botulinum toxin treatment for a long time.
4. Patients with severe mental disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of symptoms in patients with blepharospasm | up to 12 months
  Evaluation of patients with blepharospasm by rating scale.

SECONDARY OUTCOMES:
Incidence of facial numbness | up to 12 months
Incidence of facial paralysis | up to 12 months

IPD SHARING:
Plan to Share IPD: Yes